CLINICAL TRIAL: NCT06385509
Title: A Phase 4, Open-Label Study to Evaluate Primary Adrenal Function (Glucocorticoid Axis) in Hypogonadal Men Treated With JATENZO® for 12 Months
Brief Title: A Phase 4 Study to Evaluate Adrenal Function in Hypogonadal Men Treated With JATENZO® for 12 Months
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tolmar Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOL-CLAR-20024
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JATENZO® twice daily (Experimental): Participants receive 237 mg JATENZO twice daily, with the potential to be titrated to a higher or lower dose depending on serum testosterone levels.
  Interventions: Drug: Jatenzo

INTERVENTIONS:
Drug: Jatenzo — 237 mg JATENZO twice daily

SUMMARY:
TOL-CLAR-20024 is a Phase 4, multi-center, open-label safety study evaluating the potential effect of JATENZO on adrenal function in hypogonadal men treated with JATENZO for 12 months.

DETAILED DESCRIPTION:
Following all screening activities and confirmation that the subject has met all eligibility requirements, JATENZO treatment for approximately 1 year will begin. The dose of JATENZO will be titrated using its standard dose-titration algorithms based on serum testosterone levels. The Treatment Period will consist of Visits 1 - 12, with cosyntropin stimulation test completed at Visit 9 (Day 169 ±7) and Visit 12 (Day 365 ±7). At each visit during the Treatment Period, subjects will be evaluated for signs and symptoms of adrenal insufficiency, occurrence of adverse events, and changes in concomitant medications. There will be a safety follow-up visit 2 weeks after completion of Visit 12.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a man 18 to 65 years of age, inclusive, with a previous clinical diagnosis of hypogonadism (signs/symptoms consistent with hypogonadism and a low T level as defined by established criteria at the time of diagnosis); subjects must also have at least 1 T level < 300 ng/dL at either Screen 1 or Screen 2.
2. Subject must be naïve to androgen replacement therapy or washed out of prior androgen replacement therapies (wash out durations specified in exclusion criterion); that is, be willing to cease current T treatment, or currently not be taking T treatment.
3. Subject agrees as part of signed informed consent to remain off all forms of T, except for dispensed study drug, throughout the entire study.
4. Subject must have adequate venous access in the left or right arm to allow collection of blood samples.
5. Subject must be able and willing to provide written informed consent and comply with the trial protocol and procedures.

Exclusion Criteria:

* Subject will be excluded if 1 or more of the main exclusion is applicable:

  1. Subject with a history of panhypopituitarism or multiple endocrine deficiencies (whether or not on stable doses of thyroid hormone and adrenal replacement hormones).
  2. Subject with a current or prior history of AI.
  3. Subject is currently receiving corticosteroids.
  4. On the CST at Screen 3, the maximum serum total cortisol at both the 30- and 60-minute timepoint is ≤ 14 mcg/dL or has a baseline CBG outside the reference range.
  5. Subject with a history of a short course (2 weeks or less) of any glucocorticoids within the past 3 months or anabolic steroids other than testosterone within the past 6 months.
  6. Subject with a history of a protracted course of any glucocorticoid therapy (e.g., inhaled nasal steroids, inhaled oral steroids, topical steroids, injectable steroids such as joint injections) or anabolic steroids other than T. Enrolled subjects who take glucocorticoids while on study drug may be discontinued from the study at the discretion of the investigator in consultation with the sponsor.
  7. Subject with a history of anabolic steroid abuse.
  8. Subject with a diagnosis of hypogonadism who has received any topical (e.g., gel or patch), intranasal, or buccal T therapy within the previous 2 weeks, intramuscular T injection of short-acting duration (e.g., T enanthate, T cypionate) within the previous 4 weeks, intramuscular T injection of long-acting duration (e.g., AVEED®) within the previous 20 weeks, T implantable pellets (Testopel®) product within the previous 6 months or any prior use of an oral testosterone product.
  9. Subject has received any drug as part of another research study within 30 days of initial dose administration in this study.
  10. Subject has significant intercurrent disease (e.g., liver, kidney, inflammatory bowel disease, uncontrolled or poorly controlled heart disease, including hypertension, thromboembolism, congestive heart failure, or coronary heart disease, psychiatric illness, including severe depression), which in the opinion of the Investigator, would affect study participation or interpretation of study assessments.
  11. Subject has untreated, severe obstructive sleep apnea.
  12. Subject has clinically significant abnormal laboratory values, including serum transaminases > 2 × upper limits of normal (ULN), serum bilirubin > 1.5 × ULN (except subjects with Gilbert syndrome) and serum creatinine > 1.5 × ULN.
  13. Subject has a HCT value of < 35% or > 50%.
  14. Subject has a history of polycythemia, either idiopathic or associated with TRT treatment.
  15. Subject is diabetic with a glycosylated hemoglobin > 8.5%.
  16. Subject has a body mass index (BMI) ≥ 38 kg/m2.
  17. Subject has had a recent (within 2 years) history of stroke, transient ischemic attack, or acute coronary event.
  18. Subject has a mean (triplicate assessments) systolic blood pressure (sBP) > 140 mm Hg and/or diastolic blood pressure (dBP) > 90 mm Hg at screening (if prescribed antihypertensives, subject should be taking medications on the day of the screening visit with a sip of water).
  19. Subject has had recent (within 2 years) history of angina or stent (coronary or carotid) placement.
  20. Subject does not meet the requirements for concomitant medication as outlined below:

      1. If hypertensive, on a stable dose of antihypertensive medication for < 3 months
      2. If diabetic, on a stable dose of oral medication for < 2 months
      3. If on anticonvulsant therapy, on a stable dose for < 3 months
      4. If on lipid lowering medications, on a stable dose for < 3 months. Subject is expected to remain on a stable dose of lipid-lowering medication(s) throughout the study.
  21. Subject has an abnormal prostate DRE (palpable nodules), elevated PSA (serum PSA > 4.0 ng/mL), I-PSS > 19 points at screening.
  22. Subject has a history of, or current or suspected prostate cancer.
  23. Subject has a history of, or current or suspected breast cancer.
  24. Subject currently using a drug known to affect T levels, T metabolism or levels of T metabolites. These include: 5-alpha-reductase inhibitors (e.g., dutasteride, finasteride), estrogens, long-acting opioid analgesics (e.g., methadone hydrochloride, buprenorphine hydrochloride), human growth hormone (HGH) or over-the-counter supplements purported to "boost" testosterone, sexual function or improve prostate symptoms.
  25. Subject use of dietary supplements such as saw palmetto or phytoestrogens and any dietary supplements that may increase total T, such as androstenedione or dehydroepiandrosterone within the previous 4 weeks.
  26. Subject use of any over-the-counter "adrenal supplements".
  27. Subject is not willing to stop all supplemental biotin 3 days prior to testing at intervals described in this protocol.
  28. Subject currently using Megace, atypical anti-psychotics (e.g., clozapine, aripiorazole, asenapine, lumateperone, olanzapine, paliperidone, aripiprazole, ziprasidone, cariprazine, risperidone, pimavanserin, ioperidone, brexpiprazole, lurasidone, quetiapine) or chronic benzodiazepine use.
  29. Subject has a history of abnormal bleeding tendencies or thrombophlebitis unrelated to venipuncture or intravenous cannulation within the previous 2 years.
  30. Subject has history of abuse of alcohol or any drug substance within the previous 2 years.
  31. Subject deemed to be a compliance risk or unlikely to keep clinic appointments.
  32. Subject donated blood (≥ 500 mL) within the 12-week period before the initial study dose.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
CST Test | 6 months and 12 months
  To estimate the proportion of subjects with an abnormal post-stimulation cosyntropin stimulation test (CST) serum total cortisol level after approximately 6 and 12 months of treatment with JATENZO

SECONDARY OUTCOMES:
Adrenal Insufficiency | 12 months
  To estimate the proportion of subjects who develop primary adrenal insufficiency (AI) as assessed by clinical symptoms of AI and laboratory assessment of cortisol production after approximately 12 months of treatment with JATENZO

OTHER OUTCOMES:
Estrogen changes | 3 months and 6 months
  To estimate the changes from baseline in estrogen (E) after approximately 3 and 6 months of treatment with JATENZO
Follicle Stimulating Hormone (FSH) changes. | 3 months and 6 months
  To estimate the changes from baseline in follicle stimulating hormone (FSH) after approximately 3 and 6 months of treatment with JATENZO
Luteinizing hormone (LH) changes | 3 months and 6 months
  To estimate the changes from baseline in luteinizing hormone (LH) after approximately 3 and 6 months of treatment with JATENZO
Sperm analysis | 3 months and 6 months
  To estimate the changes from baseline in sperm concentration after approximately 3 and 6 months of treatment with JATENZO
Sperm analysis | 3 months and 6 months
  To estimate the changes from baseline in sperm motility after approximately 3 and 6 months of treatment with JATENZO
Sperm analysis | 3 months and 6 months
  To estimate the changes from baseline in total motile sperm count (TMSC) after approximately 3 and 6 months of treatment with JATENZO
Testis volume analysis | 3 months and 6 months
  To estimate the changes from baseline in testicular size after approximately 3 and 6 months of treatment with JATENZO

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Alliance for Multispecialty Research, Tempe, Arizona
  - Clinical Trials Research, Lincoln, California
  - Long Beach Research Institute, LLC, Long Beach, California
  - Integrated Clinical Research, Tarzana, California
  - Hillcrest Medical Research, LLC, DeLand, Florida
  - Global Health Clinical Trial Crop, Miami, Florida
  - Reserka LLC, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Velocity Clinical Research, Savannah, Georgia
  - Centennial Medical Group, Columbia, Maryland
  - Velocity Clinical Research, Omaha, Nebraska
  - AccuMed Research Associates, Garden City, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Velocity Clinical Research, Inc., Durham, North Carolina
  - Catawba Valley Medical Group, Inc., Hickory, North Carolina
  - Raleigh Medical Group, Raleigh, North Carolina
  - Piedmont Healthcare, PA, Statesville, North Carolina
  - Wilmington Health, PLLC, Wilmington, North Carolina
  - Velocity Clinical Research, Austin, Texas
  - Epic Medical Research LLC, DeSoto, Texas
  - VAST Clinical Research LLC, Garland, Texas
  - SMS Clinical Research LLC, Mesquite, Texas
  - Alpine Research Organization, Inc., Clinton, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Alliance for Multispecialty Research, Norfolk, Virginia
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No